CLINICAL TRIAL: NCT03549065
Title: Effects of Noninvasive Brain Stimulation Methods (rTMS and tDCS) Treatment on Brain Function, Craving and Relapse Prevention
Brief Title: Effects of rTMS and tDCS Treatment on Brain Function, Craving and Relapse Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: MUSouthCarolina
Record Dates: First submitted 2015-05-04; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Addiction
Keywords: Brain stimulation
MeSH Terms: conditions — Behavior, Addictive | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 20 min active tDCS, and 20 min active rTMS (Active Comparator): Applying active tDCS AND active TMS will reduce cue induced craving and opioid use, more than sham TMS AND sham tDCS and also either active TMS OR active tDCS alone. We will apply 10 daily sessions of brain stimulation (1 hour total treatment time). This is composed of 20 minutes active tDCS (anode on F3 EEG positioning and cathode on contra shoulder), followed by 4000 pulses of real rTMS (10Hz over left Dorsolateral Prefrontal Cortex(DLPFC) for 20 minutes at 120%MT). There will be 10 minutes rest between each module. We will test for cue-induced craving scores using VAS and urine drug screens for opioid abuse in comparison to the control group of sham TMS AND sham tDCS and the groups with only active tDCS OR active TMS.
  Interventions: Device: Brain Stimulation
- 20 min sham tDCS, and 20 min active rTMS (Active Comparator): Applying sham tDCS AND active TMS will reduce cue induced craving and opioid use, more than will sham TMS AND sham tDCS. We will apply 10 daily sessions of brain stimulation (1 hour total treatment time). This is composed of with 20 minutes sham tDCS (anode on F3 EEG positioning and cathode on contra shoulder), and 4000 pulses of real rTMS with (10Hz over left DLPFC for 20 minutes at 120%MT. There will be 10 minutes rest between each module. We will test for cue-induced craving scores using VAS and urine drug screens for opioid abuse in comparison to the control group of sham TMS AND sham tDCS.
  Interventions: Device: Brain Stimulation
- 20 min active tDCS, and 20 min sham rTMS (Active Comparator): Applying active tDCS AND sham TMS will reduce cue induced craving and opioid use, more than will sham TMS AND sham tDCS. We will apply 10 daily sessions of brain stimulation (1 hour total treatment time). This is composed of with 20 minutes active tDCS (anode on F3 EEG positioning and cathode on contra shoulder), and 4000 pulses of sham rTMS with (10Hz over left DLPFC for 20 minutes at 120%MT. There will be 10 minutes rest between each module. We will test for cue-induced craving scores using VAS and urine drug screens for opioid abuse in comparison to the control group of sham TMS AND sham tDCS.
  Interventions: Device: Brain Stimulation
- 20 min sham tDCS, and 20 min sham rTMS (Sham Comparator): Applying sham tDCS AND sham TMS will not reduce cue induced craving and opioid use. We will apply 10 sessions of one hour of brain stimulation. We will apply 10 daily sessions of brain stimulation (1 hour total treatment time). This is composed of with 20 minutes sham tDCS (anode on F3 EEG positioning and cathode on contra shoulder), and 4000 pulses of sham rTMS with (10Hz over left DLPFC for 20 minutes at 120%MT. There will be 10 minutes rest between each module. We will test for cue-induced craving scores using VAS and urine drug screens for opioid abuse in comparison to the control group of sham TMS AND sham tDCS.
  Interventions: Device: Brain Stimulation

INTERVENTIONS:
Device: Brain Stimulation — Transcranial magnetic stimulation (TMS) is a minimally invasive brain stimulation method that stimulates the brain of an individual focally(George & Belmaker, 2007). TMS pulses that are delivered repetitively and rhythmically are referred to as repetitive TMS (rTMS).
  Transcranial direct current stimulation (tDCS) is another form of non-invasive brain stimulation that is being investigated as an intervention for neurological and psychiatric disorders. A weak direct electrical current (0-2 mA) flows between two small electrodes via saline soaked sponges placed on the scalp (Nitsche MA et al, 2008).

SUMMARY:
Addiction is known as a chronic relapsing brain disorder that has a high cost to patients, family and society. Its ranking in cause of death is 8th globally, and substance abuse contributes 5.4% of the total global burden of disease. Brain stimulation procedures such as repetitive trans-cranial magnetic stimulation (rTMS) and trans-cranial direct current stimulation (tDCS) are considered minimal risk interventions and are used for the treatment of depression, pain, and other neurological and psychiatric disorders. There is some evidence that rTMS applied to the left prefrontal cortex results in significantly lowered craving. To date, no studies have investigated the effects of a course of either rTMS or tDCS treatment on opioid craving, brain function, and relapse prevention in opioid addicts. Individuals with prescription opioid dependence experience high rates of desire and intense cravings to use opioids. The present study aims to examine the effects of a course of daily prefrontal rTMS and tDCS on brain function, desire and craving and help to relapse prevention in abstinence phase.

DETAILED DESCRIPTION:
The investigators plan to compare and contrast TMS and tDCS alone or in combination to treat opioid abuse. We will use a 4 cell randomised parallel controlled trial, consisting of active or sham TMS, and active or sham tDCS [a-tDCS, a-TMS; s-tDCS, a-TMS; a-tDCS, s-TMS; s-tDCS, s-TMS). The investigators hypothesise that each of the active interventions alone will be superior to pure sham in reducing craving and use. Moreover, The investigators hypothesise that COMBINING the two active treatments will be synergistic and will produce the largest reductions in craving and use.

ELIGIBILITY:
Inclusion Criteria:

* 40 treatment-seeking opioid-dependent subjects (between the ages of 21 and 65) with at least 30 days of abstinence under maintenance treatment will be included in this single blind study.

Exclusion criteria includes:

* history of seizures,
* receiving any medications known to lower seizure threshold,
* pregnancy,
* metal implants above the waist,
* brain lesions or tumors,
* a history of negative reactions to TMS, and
* a positive opioid urine screen (except methadone and suboxone

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in craving and opioid relapse Using Opioid Cue panel | Day 1, 6 month
  Using Opioid Cue panel